CLINICAL TRIAL: NCT00334152
Title: A Phase III Multicenter, Randomized, Double-blind, Parallel Group Study to Evaluate the Safety and Efficacy of the 30 mg Intravenous Formulation of the Neurokinin-1 Receptor Antagonist GW679769 for Prevention of Postoperative Nausea and Vomiting in Female Subjects at High Risk for Emesis
Brief Title: Casopitant And ZOFRAN To Prevent Post Operative Nausea And Vomiting In Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NKT102552
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Nausea and Vomiting, Postoperative; Postoperative Nausea and Vomiting
Keywords: NK-1; antiemetics; casopitant mesylate; postoperative nausea and vomiting; ondansetron hydrochloride; 5HT3; ZOFRAN; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: casopitant

SUMMARY:
This study is being conducted to see if adding GW679769 (casopitant) to ZOFRAN will significantly decrease the number of patients who experience nausea and vomiting after surgery.

ELIGIBILITY:
Inclusion criteria:

* History of PONV (postoperative nausea and vomiting) and/or motion sickness.
* Have not smoked for the last 6 months.
* Having certain abdominal, breast, thyroid or shoulder surgery.

Exclusion criteria:

* Pregnant or breastfeeding.
* Have certain pre-existing medical conditions or take certain medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieved a complete response | Up to 24 hours
  Complete response defined as no vomiting or retching and no rescue therapy during the first 24 hours following placement of the last suture/staple. Vomiting defined as the forceful expulsion of gastrointestinal contents through the mouth or nose. Retching defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit that is not productive of gastrointestinal contents (also known as "dry heaves"). Study participants who receive antiemetic rescue medication(s) during the initial 24 hours was considered treatment failures.

SECONDARY OUTCOMES:
The severity of nausea experienced by participants in each cohort during the 2, 6, 24 and 48 hour periods, as assessed by an 11-point, linear, numerical rating scale referred to as a "0-10 Likert scale" | Up to 48 hours
  Nausea is defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. Each participant completed a Likert scale at 2, 6, 24 and 48 hours after placement of the last suture/staple. The Likert scale used a range of 0-10, where 0 = no nausea and 10 = nausea as bad as it could be.
The severity of nausea experienced by participants in each cohort during the 2, 6, 24 and 48 hour periods, as assessed by a categorical scale (none, mild, moderate or severe), as defined in the protocol | Up to 48 hours
  Nausea is defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. Each participant completed a categorical scale at 2, 6, 24 and 48 hours after placement of the last suture/staple. In the categorical scale, each participant asked to rate the severity of nausea as, none: no nausea, mild: queasiness/upset stomach that is manageable and minimally (if at all) affects daily activities, moderate: increased queasiness, sometimes with the feeling of having to vomit (but not vomiting), that has a significant negative effect on daily activities (for example, being unable to work, eat and drink, prepare food, care for children or others), severe: feeling sick and vomiting or feeling like you are going to vomit, and unable to perform most daily activities.
Number of participants with first emetic event | Up to 48 hours
Number of participants with first antiemetic rescue medication | Up to 48 hours
Participant satisfaction with the prophylactic antiemetic regimens, as assessed by participant satisfaction assessments in the participant diary | Up to 48 hours
Participant willingness of participants to use the same treatment regimen for future surgical procedures, as assessed by participant satisfaction assessments in the participant diary | Up to 48 hours
Number of participants with chemistry data outside the reference range | Up to 48 hours
Number of participants with hematology data outside the reference range | Up to 48 hours
Safety and tolerability of the antiemetic regimens, assessed by clinical observation (including time to awakening from anesthesia, defined as ability to respond to a verbal command) | Up to 24 hours
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Days 6-14 visit
  An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. Refer to the general AE/SAE module for a list of AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (25):
  - GSK Investigational Site, Fairhope, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Seattle, Washington
- Belgium (4):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Brasschaat
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Canada (3):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- Germany (10):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Neubrandenburg, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- Hong Kong (4):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin, New Territories
  - GSK Investigational Site, Sheung Shui, New Territories
- GSK Investigational Site, Lahore, Pakistan
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburgh
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santiago de Compostela
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKT102552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register